CLINICAL TRIAL: NCT04828213
Title: Tooth-Borne Versus Tooth-Bone-Borne Rapid Maxillary Expanders: A Stereophotogrammetric Evaluation of Soft Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gökçenur Gökçe (Other)
Responsible Party: Sponsor-Investigator, Gökçenur Gökçe, Assistant professor, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-GAP-DİŞF-0003
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Posterior Crossbite
Keywords: stereophotogrammetry; Tooth-bone-borne rapid maxillary expansion; skeletal anchorage; mini-screws

STUDY DESIGN:
Intervention Model Description: 2-arm parallel trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tooth-borne RME appliance (Hyrax) (Experimental): In the Tooth-borne RME expander group, bands were placed to the maxillary right and left upper 1st premolar and 1st molar teeth. The impression of the upper jaw was obtained with the bands in mouth by using alginate impression material. In the laboratory process, a hyrax (Forestadent, Pforzheim, Germany; Forestadent USA, St Louis, Missouri, USA) expansion appliance with an expansion screw in the middle was prepared on the models by the same technician under standard conditions.
  RME activation was performed twice a day for the first week and then once per day. When it was decided that the expansion was sufficient (until the palatal tubercles of the upper molars came into contact with the buccal tubercles of the lower molars), the screw was fixed with the 0.012-inch ligature wire (American Orthodontics) and the appliance was kept in the mouth without being activated for 3 months.
  Interventions: Device: Rapid Maxillary Expansion Treatment with Tooth-borne RME appliance (Hyrax); Device: Rapid Maxillary Expansion Treatment with Hybrid hyrax RME appliance
- Hybrid hyrax RME appliance (Experimental): Rapid Maxillary Expansion Treatment. In the Hybrid hyrax RME appliance group, mini-screws of 2 mm diameter and 9 mm length (Benefit mini-implants; PSM Medical Solutions; Tuttlingen, Germany) were placed 3 mm posterior and 1 to 5 mm paramedian to the incisive foramina.
  RME activation was performed twice a day for the first week and then once per day. When it was decided that the expansion was sufficient (until the palatal tubercles of the upper molars came into contact with the buccal tubercles of the lower molars), the screw was fixed with the 0.012-inch ligature wire (American Orthodontics) and the appliance was kept in the mouth without being activated for 3 months.
  Interventions: Device: Rapid Maxillary Expansion Treatment with Tooth-borne RME appliance (Hyrax); Device: Rapid Maxillary Expansion Treatment with Hybrid hyrax RME appliance

INTERVENTIONS:
Device: Rapid Maxillary Expansion Treatment with Tooth-borne RME appliance (Hyrax) — The patients were treated with a expansion appliance containing a Hyrax expansion screw positioned parallel to the second premolars and were used to correct the posterior crossbite. RME activation was performed twice a day for the first week and then once per day. When it was decided that the expansion was sufficient (until the palatal tubercles of the upper molars came into contact with the buccal tubercles of the lower molars), the screw was fixed with the 0.012-inch ligature wire (American Orthodontics) and the appliance was kept in the mouth without being activated for 3 months.
Device: Rapid Maxillary Expansion Treatment with Hybrid hyrax RME appliance — The patients were treated with a Hybrid hyrax RME appliance containing a Hyrax expansion screw positioned parallel to the second premolars and mini-screws. RME activation was performed twice a day for the first week and then once per day. When it was decided that the expansion was sufficient (until the palatal tubercles of the upper molars came into contact with the buccal tubercles of the lower molars), the screw was fixed with the 0.012-inch ligature wire (American Orthodontics) and the appliance was kept in the mouth without being activated for 3 months.

SUMMARY:
The force exerted by the rapid maxillary expansion (RME) appliances provides expansion of the transverse dimension by splitting of the midpalatal suture. This expansion results in three-dimensional (3D) changes in maxillary position which also effects circummaxillary surrounding structures. The aim of this randomized clinical trial (RCT) was to evaluate the effects of tooth-borne and tooth-bone-borne rapid maxillary expansion (RME) on soft tissue with stereophotogrammetry.

DETAILED DESCRIPTION:
Introduction: To evaluate the effects of tooth-borne and tooth-bone-borne rapid maxillary expansion (RME) on soft tissue with stereophotogrammetry. Methods: 32 patients (15 males, 17 females) who met inclusion criteria were divided into two groups. In the first group, tooth-borne RME appliance (Hyrax) was applied to 16 patients (9 males, 7 females mean age 13.4 ± 1.3 years) and in the second group, tooth-bone-borne RME appliance (Hybrid Hyrax) was applied to 16 patients (6 males, 10 females mean age 13.05 ±1.24 years). A simple electronically generated randomization was performed before trial commencement using the Random Allocation Software program. Allocation concealment involved numbered, sealed, and opaque envelopes prepared before trial commencement. One envelope was sequentially opened for each participant during recruitment. Each envelope contained a card with the name of 1 expander. The initials of the name of the participant, the type of expander, and the date of allocation were identified in the external surface of the envelope. One operator was responsible for the randomization process, allocation concealment, and implementation. The primary outcomes of this study was assessment of changes in soft tissues before RME (T0) and post-retention (T1) period by stereophotogrammetry. Independent and dependent sample t tests were used to compare intra- and inter-group differences at P<0.05 significance level.

ELIGIBILITY:
Inclusion Criteria:

1. No previous tonsillar, nasal or adenoid surgery and orthodontic treatment,
2. Bilateral crossbite and need for RME,
3. Maxillary and mandibular permanent teeth fully erupted,
4. Willingness to participate in the study

Exclusion Criteria:

1. the presence of adenotonsillectomy due to tonsillar hypertrophy or adenoidal hypertrophy
2. Having nasal/nasopharyngeal /oropharyngeal pathologies, craniofacial syndromes, systemic disease, poor oral hygiene,
3. History of previous orthodontic treatment.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Increasing soft tissue facial measurement-1 | At baseline and after 3 months retention period
  Increasing anterior face height
Increasing soft tissue facial measurement-2 | At baseline and after 3 months retention period
  Increasing upper lip length
Increasing soft tissue facial measurement-3 | At baseline and after 3 months retention period
  Increasing lower face height

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Akan B, Gokce G, Sahan AO, Veli I. Tooth-borne versus tooth-bone-borne rapid maxillary expanders according to a stereophotogrammetric evaluation of facial soft tissues: A randomized clinical trial. Orthod Craniofac Res. 2021 Aug;24(3):438-448. doi: 10.1111/ocr.12509. Epub 2021 Jun 21. PMID 34105880